CLINICAL TRIAL: NCT07273838
Title: Sodium-Glucose Cotransporter-2 Inhibitor for Amelioration of Acute Cardiorenal Syndrome: A Randomized Controlled Trial
Brief Title: Sodium-Glucose Cotransporter-2 Inhibitor for Patients With Acute Cardiorenal Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000038989; 1K23DK142042-01A1 (NIH)
Record Dates: First submitted 2025-08-08; First posted 2025-12-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure; Acute Kidney Injury
Keywords: Acute cardiorenal syndrome
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SGLT2i (Experimental): Subjects receive once daily 10 mg of oral dapagliflozin (Farxiga) for 14 days (or until discharge). Empaglifolozin may be used in case of dapagliflozin shortage.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Placebo (Placebo Comparator): Subjects receive once daily administration of a placebo comparator for 14 days (or until discharge).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Administration of 10mg oral dapagliflozin once daily for 14 days (or until discharge).
  Arms: SGLT2i
Drug: Placebo — Administration of placebo comparator once daily for 14 days (or until discharge).
  Arms: Placebo

SUMMARY:
The overall objective of this study is to determine whether the addition of SGLT2 inhibitors to usual care in hospitalized patients with heart failure associated acute kidney injury is safe and efficacious. Investigators will assess if SGLT2 inhibition improves a composite cardio-renal outcome (mortality, dialysis, AKI progression, decongestion metrics, heart failure symptoms). Secondary objectives of this study are to compare individual components of the composite outcome as well as changes in biomarkers of kidney injury, inflammation, repair and oxidative stress between those exposed to the SGLT2 inhibitor vs placebo.

DETAILED DESCRIPTION:
Individuals with heart failure are prone to acute kidney injury (AKI) as well as fluctuations in creatinine that meet AKI criteria. AKI diagnosis often complicates heart failure management and leads to interruptions of medications with long term benefit. AKI is also associated with long-term complications such as chronic kidney function and cardiovascular mortality. There is no efficient universal treatment for this type of AKI. In acute heart failure (AHF), although loop diuretics are the mainstay of treatment, diuretic resistance complicates the management. A drug that improves diuretic efficiency may lead to faster decongestion and improvement in kidney function.

Sodium-glucose co-transporter-2 inhibitors (SGLT2i) are drugs consistently shown to reduce hospitalizations in heart failure as well as progression of chronic kidney disease. They have also shown to promote kidney tubular health in pre-clinical models of kidney injury. They have been included in the armamentarium of heart failure care as goal directed medical therapy (GDMT) but concerns of efficacy and safety in patients with kidney dysfunction continue to limit their uptake and maintenance.

This study aims to promote increased use of SGLT2 inhibitors by demonstrating their safety and possible benefit in patients who develop kidney injury in the setting of heart failure to avoid interruptions in GDMT use.

To this end, 130 hospitalized adults with acute cardiorenal syndrome will be enrolled into a randomized controlled trial. Subjects will be randomized to receive either dapagliflozin or placebo for 14 days or until discharge (whichever comes first). Blood and urine samples will be collected for biomarker analysis, symptom and adverse event surveys will be administered, and various clinical parameters will be recorded on up to 6 study visits during hospitalization.

The primary outcome is a composite of short- and intermediate-term cardiorenal outcomes including: heart failure specific outcomes (objective measures of decongestion (i.e., effective diuresis), and a patient-reported outcome incorporating two dimensions of health state and a visual analogue scale (VAS)), kidney-specific outcomes (dialysis receipt, AKI progression to a higher stage, and change in serum creatinine), length of stay, and mortality. Secondary outcomes include trends in biomarkers of kidney injury, inflammation, oxidative stress, and repair, as well as individual components of the primary outcome as well as re-hospitalization rates.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged ≥ 18 and ≤ 85 years-old
* Diagnosed with heart failure of either preserved or reduced left ventricular function
* Have signs of heart failure exacerbation
* Ability to take an oral medication
* Willing to adhere to the SGLT2i vs placebo regimen

Exclusion Criteria:

* AKI can be primarily explained by another etiology
* Current use of SGLT2 inhibitor or exposure in the past 72 hours
* Pregnancy or lactation (pregnancy test prior to enrollment in women of child-bearing age)
* Known allergic reactions to components of an SGLT2 inhibitor
* Treatment with another investigational drug for heart failure different from or in addition to usual care within the 72 hours preceding AKI
* Any individual who meets any of the following criteria will be excluded from participation in this study:
* Documented history of ileal conduit (neobladder)
* No means of collecting urine such as patients with documented incontinence without indwelling or external urinary catheter
* Advanced kidney disease at baseline defined as baseline eGFR < 25 ml/min/1.73m2
* Unexplained hypoglycemia in the past 30 days from enrollment
* History of Fournier's gangrene (pelvic necrotizing fasciitis)
* History of recurrent urinary tract infection (UTI): defined as documented UTI at least 2x in the preceding 6 months or 3 x in the preceding 12 months
* End-stage kidney disease with dialysis requirement
* Oliguria: defined as less than 30 ml urine output per hour for more than two consecutive hours or less than 500 ml over the preceding 24 hours
* Severe acute kidney injury with indications for dialysis
* Current dialysis receipt for acute kidney injury
* Comfort measures only
* Solid organ transplant on immunosuppression

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Cardio-renal clinical improvement calculated as a Win Ratio | Calculated at 30 days post-randomization
  This outcome is assessed using a win ratio (total wins in the intervention group divided by total wins in the control group). Pairwise comparisons of predetermined components are made between each participant in the intervention and control group hierarchically in order of clinical importance, with a "win" assigned to the participant with the more favorable result at the first level of difference. The win ratio is the number of "winning" pairs for the treatment group divided by the number of "losing" pairs, with a win ratio greater than 1 indicating a benefit for the treatment.

SECONDARY OUTCOMES:
Change in slope of serum creatinine over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Measure of kidney function; assessed as a change in blood concentration.
Change in slope of serum cystatin-C over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Measure of kidney function; assessed as a change in blood concentration.
Change in slope of serum serum NT-proBNP over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Measure of kidney function; assessed as a change in blood concentration.
Change in slope of blood kidney injury molecule-1 (KIM-1) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of renal tubular injury; assessed as a change in blood concentration.
Change in slope of urine kidney injury molecule-1 (KIM-1) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of renal tubular injury; assessed as a change in urine concentration.
Change in slope of blood neutrophil gelatinase-associated lipocalin (NGAL) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of renal tubular injury; assessed as a change in blood concentration.
Change in slope of urine neutrophil gelatinase-associated lipocalin (NGAL) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of renal tubular injury; assessed as a change in urine concentration.
Change in slope of blood interleukin-6 (IL-6) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of inflammation; assessed as a change in blood concentration.
Change in slope of urine interleukin-6 (IL-6) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of inflammation; assessed as a change in urine concentration.
Change in slope of blood interluekin-18 (IL-18) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of inflammation; assessed as a change in blood concentration.
Change in slope of urine interluekin-18 (IL-18) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of inflammation; assessed as a change inurine concentration.
Change in slope of blood MPO over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of oxidative stress; assessed as a change in blood concentration.
Change in slope of urine MPO over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of oxidative stress; assessed as a change in urine concentration.
Change in slope of blood uromodulin (UMOD) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of repair; assessed as a change in blood concentration.
Change in slope of urine uromodulin (UMOD) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of repair; assessed as a change in urine concentration.
Change in slope of blood chitinase-3-like protein 1 (YKL-40) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of repair. Assessed as a change in blood concentration.
Change in slope of urine chitinase-3-like protein 1 (YKL-40) over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 +/- 4 days
  Biomarker of repair. Assessed as a change in urine concentration.
Change in slope of urine volume over 5 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4 post-enrollment
  Measure of decongestion; measured daily (i.e. every 24 hours) according to floor protocol.
Change in slope of weight over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4 and 14 post-enrollment
  Measure of decongestion; assessed upon physical exam.
Change in slope of breathlessness score over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 post-enrollment
  Measure of decongestion using a survey, scored on a Likert scale from 1-5 (5 indicates more severe breathlessness).
Change in slope of edema grade over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 post-enrollment
  Measure of decongestion; a score from 0 to 4+ is given on physical examination, with a higher score indicating higher edema.
Change in slope of patient-reported edema over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 post-enrollment
  Measure of decongestion using a survey, scored on a Likert scale from 1-5 (5 indicates more severe edema).
Change in slope of patient-reported VAS dyspnea score over 14 days from enrollment | Measured at the time of enrollment (day 0) and on days 1-4, and day 14 post-enrollment
  A patient reported outcome measured on a visual analog scale of 1-100mm, with 100 indicating worse breathlessness.
Cumulative Lasix equivalent diuretic dose over 5 days | Up to 5 days from enrollment
  Measure of decongestion
Proportion with kidney injury progression | Up to 14 days post-enrollment
  Proportion with dialysis receipt or AKI progression to a higher stage up to 14 days from enrollment
Percent survival at 30 days post-enrollment | Up to 30 days post-enrollment
  Percent of subject's surviving to 30 days post-enrollment
Percent of subjects re-hospitalized with heart failure and AKI at 30 days post-enrollment | Up to 30 days post-enrollment
  Percent of rehospitalization up to 30 days post-enrollment
Proportion with prescription of SGLT2i | Up to 30 days post-enrollment
  Proportion with prescription of SGLT2i by subject's own provider
Incidence of adverse events during exposure | Up to 14 days post-enrollment or until hospital discharge
  Number of adverse events experienced by subjects, including sodium or potassium derangements, metabolic acidosis, urinary tract infections, fungal genitourinary infection, hypotension, allergic reactions, and hypoglycemia
Change in heart failure symptoms (mobility and self care) | Measured on Days 0, 1, 2, 3, 4, and 14 post-enrollment
  Change in score using a full and modified version of the EQ-5D-5L-VAS. The full questionnaire contains 5 dimensions of state of health and the VAS (visual analog scale) addressing perceived overall health and will be conducted on day 0 and 14. The modified version contains two dimensions of health (self care and mobility) and the VAS scale, and will be conducted on days 1, 2, 3, and 4. The EQ-5D-5L dimensions are scored on a Likert Scale from 1-5, with 5 indicating worsening health. The VAS is scored on a scale of 1 to 100, with 100 indicating better perceived overall health.

CONTACTS AND LOCATIONS:
Overall Officials: Abinet Aklilu, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital-St. Raphael Campus, New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for the primary and secondary outcomes will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication; indefinitely.